CLINICAL TRIAL: NCT05477147
Title: Re-Ablation Using a Tailored Approach Targeting EGM-Dispersion
Acronym: RESTART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Volta Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLIPL-01-003
Record Dates: First submitted 2022-07-25; First posted 2022-07-28 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; AF; Artificial intelligence; Catheter Ablation; Ablation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Catheter Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Treatment Group (Experimental): Patients undergoing catheter ablation that qualify after initial screening.
  Interventions: Device: Catheter Ablation

INTERVENTIONS:
Device: Catheter Ablation — Cardiac catheter ablation for recurrent AF after previous ablation (catheter or surgical).

SUMMARY:
Multi-center, international, non-randomized clinical trial evaluating the use of Volta's VX1 algorithm as used in combination with repeat catheter ablation after AF recurrence after previous catheter ablation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 21 years of age or older indicated for redo AF ablation
2. Previous catheter or surgical ablation for paroxysmal AF, persistent AF, or long-standing persistent AF
3. Documented symptomatic AF recurrences that occurred within the last 12 months and persisted beyond 3 months after the last AF ablation procedure
4. Continuous anticoagulation with warfarin (INR 2-3) or NOAC for > 4 weeks prior to ablation
5. Patients must be able and willing to provide written informed consent to participate in the clinical trial

Exclusion Criteria:

1. Previous ablation procedure-related complication (e.g. fistula, perforation, etc.)
2. First AF ablation procedure indication was persistent AF lasting longer than 24 months
3. Long-standing persistent AF recurrence prior to study redo procedure
4. Previous AF ablation using VX1 software
5. Severe obesity (BMI > 50)
6. Very dilated Left Atrium (LA) (e.g. LA diameter > 55 mm and/or LA surface > 40 cm2 determined by 2D echocardiography)
7. Patients with AF secondary to an obvious reversible cause
8. Inadequate anticoagulation as defined in the inclusion criteria
9. LA thrombus on Transesophageal Echocardiography (TEE)* or CT Scan prior to procedure
10. Contraindications to anticoagulation (heparin, warfarin or NOAC)
11. Patients who are or may potentially be pregnant
12. Any cardiac surgery except catheter ablation within the past 2 months (60 days) (includes PCI)
13. Myocardial infarction within the past 2 months (60 days)
14. Previous AV valve surgery
15. Patient diagnosed with hypertrophic cardiomyopathy
16. History of blood clotting or bleeding abnormalities
17. Documented arterial thromboembolic event (including TIA) within the past 12 months (365 days)
18. Rheumatic Heart Disease
19. Cardiac Sarcoidosis
20. Chronic severe Heart Failure (NYHA functional class IV and/or LVEF < 25%)
21. Awaiting cardiac transplantation or other cardiac surgery within the next 12 months (365 days)
22. Unstable angina within the past month
23. Acute illness or active systemic infection or sepsis
24. AF secondary to electrolyte imbalance, thyroid disease, or reversible or non-cardiac cause
25. Diagnosed atrial myxoma
26. Significant severe pulmonary disease (e.g. patients with restrictive pulmonary disease, constrictive or chronic obstructive pulmonary disease in GOLD stage IV) or any other disease or malfunction of the lungs or respiratory system that produces chronic symptoms (e.g. unstable or untreated sleep apnea)
27. Significant congenital anomaly or medical problem that in the opinion of the investigator would preclude enrollment
28. Enrollment in an investigational study evaluating another device, biologic, or drug
29. Presence of intramural thrombus, tumor or other abnormality or condition that precludes vascular access, or manipulation of the catheter
30. Life expectancy or other disease processes likely to limit survival to less than 12 months
31. Acute Covid-19 infection (fever and/or biological inflammatory syndrome, and positive test documented)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2023-03-17 (Actual); Primary Completion 2025-05-07 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Freedom from AF | 1 year
  Percent of patient free from recurrent AF episodes of >30 seconds at 1 year after 1 study redo procedure

CONTACTS AND LOCATIONS:
Locations (19):
- United States (15):
  - Grandview Medical Center, Birmingham, Alabama
  - Arrhythmia Research Group, Jonesboro, Arkansas
  - Ascension St. Vincent's Hospital, Jacksonville, Florida
  - Northshore University Health System, Evanston, Illinois
  - Northwestern University, Evanston, Illinois
  - Loyola University, Maywood, Illinois
  - Kansas City Cardiac Arrhythmia Research LLC, Overland Park, Kansas
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Washington University, St Louis, Missouri
  - Northwell Health System, New York, New York
  - The Ohio State University, Columbus, Ohio
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - Allegheny Health Network, Pittsburgh, Pennsylvania
  - Houston Methodist Research Institute, Houston, Texas
  - Inova Fairfax Hospital, Fairfax, Virginia
- OLV Aalst, Aalst, Belgium
- France (2):
  - Hôpital Privé Jacques Cartier, Massy
  - Clinique Pasteur, Toulouse
- Deutsches Herzzentrum München, München, Germany

IPD SHARING:
Plan to Share IPD: No